CLINICAL TRIAL: NCT02496052
Title: The Efficacy and Safety of the Dried Biological Amnion Graft Following Hysteroscopic Lysis for the Prevention of Postoperative Adhesions in Patients With Intrauterine Adhesions
Brief Title: The Efficacy and Safety of the Dried Biological Amnion Graft in Patients With Intrauterine Adhesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Obstetrics and Gynecology Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NO.1-20140601; 2014-1-2112 (Other Grant/Funding Number: The capital health research and development of special); zylx201406 (Other Grant/Funding Number: Beijing Municipal Administration of Hospitals Clinical Medicine Development of Special Funding Support)
Record Dates: First submitted 2015-07-06; First posted 2015-07-14 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Intrauterine Adhesions
Keywords: amnion graft; New biological barrier system
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- dried biological amnion graft (Experimental): patients, who are with IUA, treated by uterine application of amnion membrane + Foley balloon+ hormones (estradiol valerate tablets+dydrogesterone Tablets) following hysteroscopic adhesiolysis.
  Interventions: Procedure: dried biological amnion graft; Device: Foley balloon; Drug: estradiol valerate tablets+dydrogesterone Tablets
- Foley catheter balloon only (Sham Comparator): patients, who are with IUA, treated by uterine application of Foley balloon only+ hormones (estradiol valerate tablets+dydrogesterone Tablets) following hysteroscopic adhesiolysis.
  Interventions: Device: Foley balloon; Drug: estradiol valerate tablets+dydrogesterone Tablets

INTERVENTIONS:
Procedure: dried biological amnion graft — Uterine application of amnion membrane following hysteroscopic adhesiolysis. Other Name: Human amnion membrane
  Other Names: Uterine application of amnion membrane
  Arms: dried biological amnion graft
Device: Foley balloon — Device: Foley balloon Uterine application of Foley balloon
  Other Names: Device: Foley balloon Uterine application of Foley balloon
Drug: estradiol valerate tablets+dydrogesterone Tablets — oral estradiol valerate tablets+dydrogesterone Tablets
  Other Names: Progynova+dydrogesterone

SUMMARY:
To estimate the efficacy and safety of dried biological amnion graft after hysteroscopic lysis of intrauterine adhesions.

DETAILED DESCRIPTION:
Allocation: Randomized Endpoint Classification: Safety/Efficacy Study Intervention Model: Parallel Assignment Masking: Single Blind (Subject) Primary Purpose: Prevention

ELIGIBILITY:
Inclusion Criteria:

* age 20-40 years；
* previously diagnostic hysteroscopy confirmed adhesion score >5， according to the American Fertility Society （AFS）classification of IUA；
* complains of menstruation disorder and reproductive dysfunction；
* informed consent.

Exclusion Criteria:

* premature menopause,
* presence of other intrauterine lesions (e.g. polyps, myoma, septa), and
* presence of severe intercurrent illness (e.g. systemic disease, coagulative disorders, severe kidney and liver diseases),
* adhesions limited to the lower uterine cavity or the cervical canal.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
second diagnostic hysteroscopy | postoperation three to four months

CONTACTS AND LOCATIONS:
Overall Officials: Duan Hua, Ph.D, Study Chair — Beijing Obstetrics and Gynecology Hospital
Locations (1):
- Beijing Obstetrics and Gynecology Hospital，Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Amer MI, Abd-El-Maeboud KH. Amnion graft following hysteroscopic lysis of intrauterine adhesions. J Obstet Gynaecol Res. 2006 Dec;32(6):559-66. doi: 10.1111/j.1447-0756.2006.00454.x. PMID 17100817
- [Derived] Gan L, Duan H, Sun FQ, Xu Q, Tang YQ, Wang S. Efficacy of freeze-dried amnion graft following hysteroscopic adhesiolysis of severe intrauterine adhesions. Int J Gynaecol Obstet. 2017 May;137(2):116-122. doi: 10.1002/ijgo.12112. Epub 2017 Mar 1. PMID 28170094